CLINICAL TRIAL: NCT01671579
Title: Comparison of Bowel Ultrasound & MR Enterography in the Follow-up of Previously Diagnosed Pediatric Sm. Bowel Crohn Disease.
Brief Title: Comparison of Bowel Ultrasound & MR Enterography in the Follow-up of Previously Diagnosed Pediatric Small Bowel Crohn Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI changed institutions
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Jonathan Dillman, MD, Principal Investigator, Children's Hospital Medical Center, Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00061688
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pediatric small bowel Crohn disease (Other): Subjects with previously diagnosed PSBCD (pediatric small bowel Crohn disease)who are scheduled for a clinically MRE (magnetic resonance enterography)imaging exam.
  Interventions: Procedure: Bowel ultrasound; Procedure: magnetic resonance enterography (MRE)

INTERVENTIONS:
Procedure: Bowel ultrasound — The ultrasound imaging will take place prior to the clinically ordered MRE exam. The subject will be asked to lie on the ultrasound table for approximately 60 minutes while a variety of ultrasound images are completed.
  Other Names: abdominal ultrasound imaging; ultrasound elasticity imaging
Procedure: magnetic resonance enterography (MRE) — The subject will have a small intravenous (IV) catheter placed in on of their arms before the MRE exam. Medications called Glucagon and MultiHance will be given thru the IV catheter during the imaging study. The glucagon will decrease the movement of the intestines, which helps provide better images of the bowel. MultiHance is a contrast that helps create clearer MRE images. In addition to the MultiHance, the subject will be given an oral contrast medication called VoLumen to drink approximately 45 minutes before the MRE imaging is started. These medications are used for all clinically necessary MRE studies performed in children and adults at the UMHS. The MRE will take approximately 50 to 60 minutes to complete.

SUMMARY:
To establish the accuracy of bowel ultrasound in the follow-up of known (previously diagnosed) pediatric small bowel Crohn disease, using MR Enterography (magnetic resonance imaging technology used to obtain detailed images of the small bowel) as the reference standard.

DETAILED DESCRIPTION:
25-30% of individuals with Crohn disease present during childhood or adolescence, and the incidence is rising. MRE (magnetic resonance enterography) is considered the standard of care for imaging of pediatric small bowel Crohn's disease. Bowel ultrasound is an emerging technology for bowel assessment and offers several advantages over MRE, including lower cost, shorter exam time, and lack of need for sedation and contrast materials and bowel medication. The researchers goal is to assess the accuracy of bowel ultrasound in the follow-up of known pediatric small bowel Crohn disease using MRE and the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or younger
* Subjects with known small bowel Crohn disease undergoing a clinically ordered imaging follow-up with MR enterography.

Exclusion Criteria:

* Subjects with suspected or newly diagnosed Crohn disease
* Subject who have the following in their body may not undergo MRE imaging:

  * Metal chips/shrapnel
  * Surgical clips
  * Artificial joints
  * Metallic bone plates
  * Prosthetic devices
  * Heart pacemakers
  * Clips in or around the eye balls
  * artificial heart valves
  * Bullet fragments
  * Chemotherapy or insulin pumps

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2012-03; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Follow-up of known small bowel Crohn disease | 1 year
  A variety of imaging findings will be documented by ultrasound and correlated with the imaging findings from the clinically ordered MRE exam to determine the efficacy of bowel ultrasound in the follow-up of small bowel Crohn disease in pediatric subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R. Dillman, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States